CLINICAL TRIAL: NCT05233644
Title: Study Title Medikamentenadhärenz Bei Erwachsenen Personen Mit Herzinsuffizienz
Brief Title: Medication Adherence in Heart Failure After Hospitalisation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01733
Record Dates: First submitted 2021-10-28; First posted 2022-02-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Adherence, Medication; Heart Failure
MeSH Terms: conditions — Medication Adherence; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore medication adherence in patients who were hospitalised due to heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart failure
* Hospitalisation due to heart failure in the past two years

Exclusion Criteria:

* Not speaking German
* cognitive impairment

Min Age: 118 Years | Sex: All
Age Groups: Older Adult
Study Population: Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | at one timepoint (cross sectional)
  MARS-5 5-Item Medication Adherence Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided